CLINICAL TRIAL: NCT04005924
Title: An Acute, Randomized, Double-blind, Controlled, Crossover Study to Investigate the Effect of an Arabinogalactan Product on Glucose and Insulin Response in Adults
Brief Title: Effect of an Arabinogalactan Product
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biofortis, Merieux NutriSciences (Industry)
Collaborators: Lonza Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: BIO 1904
Record Dates: First submitted 2019-06-27; First posted 2019-07-02 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Postprandial Blood Glucose
Keywords: blood glucose; blood insulin; postprandial; fiber
MeSH Terms: interventions — arabinogalactan; Bread; Junctional Adhesion Molecule A

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Bread and sugar-free blackberry jam breakfast
- Low dose (Experimental): Bread and sugar-free blackberry jam breakfast with 6 g arabinogalactan
  Interventions: Other: arabinogalactan
- High dose (Experimental): Bread and sugar-free blackberry jam breakfast with 21 g arabinogalactan
  Interventions: Other: arabinogalactan

INTERVENTIONS:
Other: arabinogalactan — Arabinogalactan will be mixed into sugar-free blackberry jam and consumed with the provided bread.
  Other Names: control breakfast; bread plus jam
  Arms: High dose; Low dose

SUMMARY:
Dietary fiber is an important nutrient that supports gastrointestinal function as well as blood glucose and cholesterol maintenance. The National Academy of Sciences Institute of Medicine (IOM) established an adequate intake for fiber as 14 g/kcal, or 38 g and 25 g for men and women, respectively. Currently, however, the majority of the U.S. population falls substantially below this level, with mean intakes of 18.9 g/day and 15.7 g/day in men and women age 20 and older, respectively. Fiber is a complex category that contains a number of different polysaccharides and oligosaccharides that are not digested in the upper gastrointestinal tract. In its final rule updating the Nutrition and Supplement Facts label regulations, which was published in May 2016, the U.S. FDA revised the definition of dietary fiber for food labeling and included two categories: (1) the intrinsic and intact non-digestible carbohydrate (NDC) and lignin, and (2) the isolated or synthesized NDC. In this re-definition, those NDCs that are isolated from plant and other food sources will now require clinical data indicating that the ingredient provides a physiological effect that is beneficial to human health.

This study is designed to test the effect of an isolated NDC, arabinogalactan, on attenuation of blood glucose and/or insulin. Attenuation of blood glucose and/or insulin is one of the outcomes identified by the U.S. FDA as a physiological effect that is beneficial to human health, and as such, can be used to support that an isolated NDC is acting as a fiber (FDA 2018). Arabinogalactans are hemicelluloses that are abundant in plants. Arabinogalactans are found in seeds, leaves, roots, and fruit of higher plants, such as cereals, beans, leeks, pear, corn, and wheat (Saeed 2011; Dion 2016). The arabinogalactan ingredient used in the study is isolated from larch (Larix laricina) using a patented water-based extraction process. Larch arabinogalactan has been designated as Generally Recognized as Safe (GRAS) by the U.S. FDA (2000) for multiple uses and has been used in numerous previous clinical studies in humans, with no significant safety issues observed at intakes of up to 30 g daily for up to 6 weeks. The present study was designed with the goal to assess the effect of acute consumption of arabinogalactan on blood glucose and insulin responses.

DETAILED DESCRIPTION:
The study is an acute, single-center, randomized, controlled, crossover trial with one screening visit (Visit 1; Day -7) and 3 test visits (Visits 2, 3, and 4; Days 0, 7, and 14). The three test visits are each separated by a 7-day washout period.

At Visit 1 (Day -7), subjects will provide informed consent and a fasting capillary blood glucose will be assessed for eligibility purposes (fasting blood glucose must be ≥70 mg/dL and ≤125 mg/dL). At Visit 1, the following will also be conducted: medical history and prior and current medication/supplement use, inclusion and exclusion criteria, and vein access (using the Vein Access Scale; Appendix 2) will be assessed; and height, body weight, and vital signs will be measured; and BMI will be calculated. Fasting (12 ± 2 h) blood samples will be collected for chemistry and hematology, and female subjects <60 years old will undergo an in-clinic urine pregnancy test. Prior to release from the clinic, all subjects will be provided study instructions to follow before the next visit, which include: maintenance of adequate hydration and habitual diet/physical activity (throughout the study); fasting (12 ± 2 h, water only, prior to test visits); consumption of a diet that incorporates at least 150 g of total carbohydrate, refraining from vigorous physical activity (i.e., sweat-inducing exercise), and alcohol consumption (24 h prior to test visits); and refraining from tobacco (1 h before and during test visits). Subjects will then be dispensed a 24-h Diet Record with instructions to record all food and beverage intake the day prior to the first test visit (Visit 2, Day 0) and released from the clinic.

At Visit 2 (Day 0), subjects will arrive at the clinic fasted (12 ± 2 h, water only) to undergo clinic visit procedures (assessment for concomitant medication/supplement use, body weight, and vital signs). Eligible subjects will then be formally entered into the testing phase of the trial and assigned to a random test sequence. Adverse events (AE) will be assessed and subjects will be queried about compliance with study and test day instructions. Additionally, the 24-h Diet Record will be collected and reviewed. Subjects will undergo the glycemic/insulinemic response test with blood glucose concentrations obtained via capillary measurement and insulin concentrations assessed via venous measurement. An intravenous catheter will be inserted at least 10 min prior to the first blood sampling time. In order to maintain patency of the intravenous catheter, the catheter will be flushed with normal saline solution at least hourly. Blood samples will be drawn by venipuncture if the catheter fails.

Baseline capillary and venous blood samples will be collected at t= -15 and -5 min prior to beginning the meal consumption. Subjects will be instructed to begin consumption of the breakfast meal at t = 0 min and required to consume the meal in its entirety within 10 min. Capillary and venous blood samples will then be obtained at t = 15, 30, 45, 60, 75, 90, and 120 ± 5 min, where t=0 is the start of breakfast meal consumption. Additional venous blood samples will be collected as back-ups at all time points. Following the last blood draw, AEs will be assessed and subjects will begin their 7-day washout. Subjects will be dispensed a blank 24-h Diet Record with instructions to record intake the day prior to each test visit (i.e., Visits 3 and 4 (Days 7 and 14) and a copy of their first 24-h Diet Record with instructions to replicate their diet to the best of their abilities the day prior to each test visit (i.e., Visits 3 and 4 (Days 7 and 14). Subjects will also be reminded of the study instructions as per Visit 1, Day -7 (see above).

At Visits 3 and 4 (Day 7 and 14), subjects will return to the clinic, crossover to the next study breakfast meal in their respective test sequence, and repeat the procedures from Visit 2 (Day 0).

ELIGIBILITY:
Inclusion Criteria:

1. Subject is a male or female, 21-65 years of age, inclusive at Visit 1 (Day -7).
2. Subject has a BMI of 18.5 to 32.0 kg/m2, inclusive, at Visit 1 (Day -7).
3. Subject has a rating of 7 to 10 on the Vein Access Scale at Visit 1 (Day -7; Appendix 2).
4. Subject has no plans to change smoking habits during the study period and is able to abstain from tobacco products 1 h prior to and during each test visit (Visits 2, 3, and 4; Days 0, 7 and 14).
5. Subject is willing to maintain physical activity patterns, body weight, and habitual diet throughout the trial.
6. Subject is willing to abstain from alcohol consumption and avoid vigorous physical activity for 24 h prior to all test visits (Visits 2, 3, and 4; Days 0, 7, and 14).
7. Subject has no health conditions that would prevent him/her from fulfilling the study requirements as judged by the Clinical Investigator on the basis of medical history and routine laboratory test results.
8. Subject understands the study procedures and signs forms providing informed consent to participate in the study and authorizes the release of relevant protected health information to the Clinical Investigator.

Exclusion Criteria:

1. Subject has diagnosed diabetes mellitus (Type 1 or Type 2) or fasting glucose >125 mg/dL at Visit 1 (Day -7).
2. Subject has a fasting glucose <70 mg/dL at Visit 1 (Day -7).
3. Subject has a history or presence of uncontrolled and/or clinically important pulmonary (including uncontrolled asthma), cardiac (including, but not limited to, atherosclerotic disease, history of myocardial infarction, peripheral arterial disease, stroke), hepatic, renal, gastrointestinal (including but not limited to inflammatory bowel diseases, such as Crohn's disease and ulcerative colitis, celiac disease), endocrine, hematologic, immunologic, neurologic (such as Alzheimer's or Parkinson's disease), psychiatric (including depression and/or anxiety disorders) or biliary disorders.
4. Subject has a known allergy (e.g. gluten allergy), intolerance (e.g. gluten intolerance), or sensitivity to any of the foods or ingredients in the study meals.
5. Subject has extreme dietary habits (e.g., Atkins diet/ketogenic, very high protein, very high fiber, vegetarian), in the opinion of the Clinical Investigator.
6. Subject has uncontrolled hypertension (systolic blood pressure ≥140 mm Hg or diastolic blood pressure ≥90 mm Hg) as defined by the blood pressure measured at Visit 1 (Day -7). One re-test will be allowed on a separate day prior to Visit 2 (Day 0), for subjects whose blood pressure exceeds either of these cut points at Visit 1 (Day -7), in the judgment of the Clinical Investigator.
7. Subject has a history or presence of cancer in the prior 2 years, except for non-melanoma skin cancer.
8. Subject has a history of bariatric surgery for weight reducing purposes.
9. Subject has experienced any major trauma or any other surgical event within 3 months of Visit 1 (Day -7).
10. Subject has had a weight loss or gain >4.5 kg in the 3 months prior to Visit 1 (Day -7).
11. Subject has used any over-the-counter or prescription medications [with the exception of contraceptives, stable dose (defined as 90 days prior to Visit 1) statins and anti-hypertensive medications] and/or dietary supplements (other than a standard multivitamin/mineral supplement) within 3 weeks of Visit 1 (Day -7).
12. Subject has any signs or symptoms of an active infection of clinical relevance (e.g., urinary tract or respiratory) within 5 days prior to Visit 1.
13. Subject has been exposed to any non-registered drug product within 30 days prior to Visit 1 (Day -7).
14. Subject is a heavy smoker (defined as 1 pack/day of cigarettes) and/or user of marijuana products or products that contain cannabinoids.
15. Subject has a recent history of (within 12 months of screening; Visit 1; Day -7) or strong potential for alcohol or substance abuse. Alcohol abuse is defined as >14 drinks per week (1 drink = 12 oz beer, 5 oz wine, or 1½ oz distilled spirits).
16. Subject has a condition the Clinical Investigator believes would interfere with his ability to provide informed consent, comply with the study protocol, which might confound the interpretation of the study results, or put the subject at undue risk.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-05-06 (Actual); Primary Completion 2019-08-19 (Actual); Study Completion 2019-10-08 (Actual)

PRIMARY OUTCOMES:
iAUC of blood glucose | Blood glucose will be determined at 8 time points, including immediately prior to the consumption of breakfast and up to 2 hours post consumption, during 3 study visits.
  Difference in 2-h incremental area under the curve (iAUC) for postprandial blood glucose between test breakfasts with arabinogalactan and control.

SECONDARY OUTCOMES:
Cmax of blood glucose | Cmax will be obtained during 3 study visits. Blood glucose will be determined at 8 time points including immediately prior to the consumption of breakfast and up to 2 hours post consumption.
  Maximum concentration (Cmax) for postprandial blood glucose during each study visit
iAUC of blood insulin | Blood insulin will be determined at the same 8 time points as blood glucose during 3 study visits.
  Difference in 2-h incremental area under the curve (iAUC) for postprandial blood insulin between test breakfasts with arabinogalactan and control.
Cmax of blood insulin | Cmax will be obtained during 3 study visits. Blood insulin will be determined at 8 time points including immediately prior to the consumption of breakfast and up to 2 hours post consumption.
  the largest postprandial blood insulin concentration during each study visit
Tmax of blood glucose | Tmax will be obtained during 3 study visits. Blood glucose will be determined at 8 time points including immediately prior to the consumption of breakfast and up to 2 hours post consumption.
  Time to reach Cmax of blood glucose during each study visit
Tmax of blood insulin | Tmax will be obtained during 3 study visits. Blood insulin will be determined at 8 time points including immediately prior to the consumption of breakfast and up to 2 hours post consumption.
  Time to reach Cmax of blood insulin during each study visit

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Lawless, MD, Principal Investigator — Biofortis, Merieux NutriSciences
Locations (1):
- Oliver Chen, Addison, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dion C, Chappuis E, Ripoll C. Does larch arabinogalactan enhance immune function? A review of mechanistic and clinical trials. Nutr Metab (Lond). 2016 Apr 12;13:28. doi: 10.1186/s12986-016-0086-x. eCollection 2016. PMID 27073407
- [Background] Garcia AL, Otto B, Reich SC, Weickert MO, Steiniger J, Machowetz A, Rudovich NN, Mohlig M, Katz N, Speth M, Meuser F, Doerfer J, Zunft HJ, Pfeiffer AH, Koebnick C. Arabinoxylan consumption decreases postprandial serum glucose, serum insulin and plasma total ghrelin response in subjects with impaired glucose tolerance. Eur J Clin Nutr. 2007 Mar;61(3):334-41. doi: 10.1038/sj.ejcn.1602525. Epub 2006 Sep 20. PMID 16988651
- [Background] Garcia AL, Steiniger J, Reich SC, Weickert MO, Harsch I, Machowetz A, Mohlig M, Spranger J, Rudovich NN, Meuser F, Doerfer J, Katz N, Speth M, Zunft HJ, Pfeiffer AH, Koebnick C. Arabinoxylan fibre consumption improved glucose metabolism, but did not affect serum adipokines in subjects with impaired glucose tolerance. Horm Metab Res. 2006 Nov;38(11):761-6. doi: 10.1055/s-2006-955089. PMID 17111305
- [Background] Hartvigsen ML, Laerke HN, Overgaard A, Holst JJ, Bach Knudsen KE, Hermansen K. Postprandial effects of test meals including concentrated arabinoxylan and whole grain rye in subjects with the metabolic syndrome: a randomised study. Eur J Clin Nutr. 2014 May;68(5):567-74. doi: 10.1038/ejcn.2014.25. Epub 2014 Mar 5. PMID 24595224
- [Background] Hartvigsen ML, Gregersen S, Laerke HN, Holst JJ, Bach Knudsen KE, Hermansen K. Effects of concentrated arabinoxylan and beta-glucan compared with refined wheat and whole grain rye on glucose and appetite in subjects with the metabolic syndrome: a randomized study. Eur J Clin Nutr. 2014 Jan;68(1):84-90. doi: 10.1038/ejcn.2013.236. Epub 2013 Nov 20. PMID 24253758
- [Background] Lu ZX, Walker KZ, Muir JG, Mascara T, O'Dea K. Arabinoxylan fiber, a byproduct of wheat flour processing, reduces the postprandial glucose response in normoglycemic subjects. Am J Clin Nutr. 2000 May;71(5):1123-8. doi: 10.1093/ajcn/71.5.1123. PMID 10799374
- [Background] Robinson RR, Feirtag J, Slavin JL. Effects of dietary arabinogalactan on gastrointestinal and blood parameters in healthy human subjects. J Am Coll Nutr. 2001 Aug;20(4):279-85. doi: 10.1080/07315724.2001.10719048. PMID 11506055
- [Background] Saeed F, Pasha I, Anjum FM, Sultan MT. Arabinoxylans and arabinogalactans: a comprehensive treatise. Crit Rev Food Sci Nutr. 2011 May;51(5):467-76. doi: 10.1080/10408391003681418. PMID 21491271
- See also: Scientific evaluation of the evidence on the beneficial physiological effects of isolated or synthetic non-digestible carbohydrates submitted as a Citizen Petition (21 CFR 10.30): Guidance for Industry. — https://www.fda.gov/regulatory-information/search-fda-guidance-documents/guidance-industry-scientific-evaluation-evidence-beneficial-physiological-effects-isolated-or
- See also: What We Eat in America, NHANES 2015-2016. — https://www.ars.usda.gov/ARSUserFiles/80400530/pdf/1516/Table_1_NIN_GEN_15.pdf